CLINICAL TRIAL: NCT00004064
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase IIB Study of the Safety and Efficacy of OVAREX MabB43.13 in Ovarian Cancer Patients With an Elevated Serum CA 125 But Without Other Evidence of Disease
Brief Title: Monoclonal Antibody Therapy in Treating Patients With Ovarian, Fallopian Tube, or Peritoneal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: AltaRex (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000067265; ALTAREX-OVA-Gy-10; OU-08111
Record Dates: First submitted 1999-12-10; First posted 2004-08-05 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2007-06

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: stage I ovarian epithelial cancer; stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; fallopian tube cancer; primary peritoneal cavity cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — oregovomab

INTERVENTIONS:
Biological: oregovomab

SUMMARY:
RATIONALE: Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells.

PURPOSE: Randomized phase II trial to study the effectiveness of monoclonal antibody therapy in treating patients who have ovarian, fallopian tube, or peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the safety of OvaRex monoclonal antibody B43.13 in patients with elevated CA 125 and histologically proven epithelial adenocarcinoma of the ovary, fallopian tube, or peritoneum, but without other evidence of disease. II. Determine the time to disease progression, overall survival, CA 125 levels, immune responses, and quality of life of these patients treated with this regimen.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 2 treatment arms: Arm I: Patients receive placebo IV during weeks 1, 3, 5, 9, 13, 25, 37, and 49. Arm II: Patients receive OvaRex monoclonal antibody B43.13 (MOAB B43.13) IV during weeks 1, 3, 5, 9, 13, 25, 37, and 49. Patients in either treatment arm who have no disease progression after week 49 receive MOAB B43.13 once every 12 weeks until week 121. Patients with disease progression after week 49 may receive MOAB B43.13 alone, in combination with, or following chemotherapy. Quality of life is assessed during the study.

PROJECTED ACCRUAL: A total of 102 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven epithelial adenocarcinoma of the ovary, fallopian tube, or peritoneum CA 125 greater than 35 U/mL No conclusive radiological or clinical evidence of disease No disease recurrence Must have received only 1 prior platinum based chemotherapy regimen No tumors of low malignant potential or noninvasive disease

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 6 months Hematopoietic: Hemoglobin at least 8.0 g/dL Lymphocyte count at least 1,000/mm3 Neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 times normal Renal: Creatinine no greater than 2 mg/dL Cardiovascular: No uncontrolled hypertension No congestive heart failure No arrhythmias Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No active autoimmune disease requiring chronic treatment No allergy to murine proteins No documented anaphylactic reaction to any drug No active infection causing fever No immunodeficiency disease No uncontrolled nonmalignant diseases No other malignancy (except nonmelanomatous skin cancer or carcinoma in situ of the cervix) unless curatively treated and free of disease for at least 5 years

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior murine monoclonal antibodies Chemotherapy: See Disease Characteristics At least 4 weeks since prior platinum based chemotherapy No concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: At least 6 months since prior limited field (i.e., abdominal or pelvic) radiotherapy No prior whole abdominal radiotherapy Surgery: At least 4 weeks since prior surgery No prior splenectomy Other: At least 4 weeks since prior immunosuppressive drugs No concurrent immunosuppressive drugs At least 30 days since other prior investigational drugs

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 1998-11

CONTACTS AND LOCATIONS:
Overall Officials: Michael A. Bookman, MD, Study Chair — Fox Chase Cancer Center
Locations (16):
- United States (15):
  - Gynecologic Oncology Associates, Newport Beach, California
  - Lee Memorial Health System, Fort Myers, Florida
  - Walt Disney Memorial Cancer Institute, Orlando, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Indiana University Cancer Center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Mercy Medical Center, Inc., Baltimore, Maryland
  - Barnes-Jewish Hospital, St Louis, Missouri
  - St. John's Mercy Medical Center, St Louis, Missouri
  - University of Oklahoma College of Medicine, Oklahoma City, Oklahoma
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Palmetto Richland Memorial Hospital, Columbia, South Carolina
  - Texas Oncology, P.A., Dallas, Texas
  - Cancer Center, University of Virginia HSC, Charlottesville, Virginia
  - Riverside Regional Medical Center, Newport News, Virginia
- Ottawa Regional Cancer Center - General Division, Ottawa, Ontario, Canada